CLINICAL TRIAL: NCT02744976
Title: Coronary Artery Disease Progression by iMap Intravascular Ultrasound Analysis in Patients With Prediabetes
Brief Title: Coronary Artery Disease Progression in Patients With Prediabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pauls Stradins Clinical University Hospital (Other)
Responsible Party: Principal Investigator, Karlis Trusinskis, MD, PhD, Pauls Stradins Clinical University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IVUS-0216
Record Dates: First submitted 2016-04-15; First posted 2016-04-20 (Estimated); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Coronary Artery Disease; Atherosclerosis; Prediabetic State
Keywords: Coronary artery disease; Atherosclerosis; Prediabetes; Intravascular ultrasound; Insulin resistance; Percutaneous coronary intervention; Metformin
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Prediabetic State; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prediabetes, metformin (Experimental): Patients with HbA1c 5.7-6.4 receiving metformin and lifestyle recommendations
  Interventions: Drug: Metformin; Behavioral: Lifestyle recommendations
- Prediabetes, lifestyle (Active Comparator): Patients with HbA1c 5.7-6.4 receiving lifestyle recommendations
  Interventions: Behavioral: Lifestyle recommendations

INTERVENTIONS:
Drug: Metformin — In order to minimize gastrointestinal discomfort, metformin treatment will be started with a dose of 500 mg p/o once daily, then gradually increased to 2000 mg p/o once daily for 24 months
  Other Names: Glucophage extended release (XR)
  Arms: Prediabetes, metformin
Behavioral: Lifestyle recommendations — Standard lifestyle recommendations

SUMMARY:
Prediabetes is a disorder of glucose metabolism that reflects the natural history of progression from normoglycaemia to type 2 diabetes mellitus. Patients with prediabetes have impaired glucose regulation caused by insulin resistance (IR). IR in patients undergoing percutaneous coronary intervention (PCI) is associated with coronary artery remodeling and coronary plaque vulnerability by intravascular ultrasound (IVUS) analysis. In stent restenosis after bare metal and drug-eluting stent implantation more frequently is observed in patients with high fasting-insulin levels and IR. Although IR has a significant role in the progression of atherosclerosis in prediabetic patients, the importance of managing prediabetes is often under-appreciated by clinicians. To date, no pharmacological treatment has been officially approved for prediabetes. According to American Diabetes Association recommendations, metformin is the only drug that could be considered in the treatment of prediabetic patients with a high risk of developing diabetes. Metformin is a safe and inexpensive glucose lowering drug that attenuates mortality and future cardiovascular events in patients with type 2 diabetes as well as the progression of atherosclerosis in non-diabetic animal models. This study was designed to analyze coronary plaque characteristics by iMAP IVUS in patients with and without prediabetes undergoing PCI and to evaluate the impact of metformin treatment on coronary plaque characteristics in prediabetic patients at 24 month follow up.

The study hypothesis is that more pronounced coronary atherosclerosis progression as well as in-stent neointimal hyperplasia will be observed in patients with prediabetes. Metformin treatment attenuates the progression of atherosclerosis in patients with prediabetes.

DETAILED DESCRIPTION:
Patients undergoing PCI and IVUS pullback for the target vessel will be enrolled in a prospective study. Before PCI and at 24 month follow up fasting blood will be collected for glucose, HbA1c, C peptide, lipid profile assessment. Patients' baseline demographic characteristics, medical history, and procedural data will be collected during the index hospitalization and at 24 month follow up. Patients will be divided in groups according to HbA1c - control group (HbA1c<5.7) and prediabetic patients (HbA1c 5.7-6.4). PCI will be performed in accordance with the guidelines. After successful treatment of the culprit lesion IVUS will be done. Following PCI and IVUS patients with prediabetes will be randomly assigned in groups either receiving metformin at a dose of 2000 mg once daily plus standard lifestyle recommendations or standard lifestyle recommendations only. Intravascular ultrasound analysis will be repeated 24 months after the initial PCI.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 and <75 years;
* patients with stable coronary artery disease referred to PCI in an artery suitable for IVUS pullback;
* signed informed consent before PCI.

Exclusion Criteria:

* cardiac or non-cardiac illness with life expectancy of less than two years;
* failure to advance the IVUS catheter through the culprit lesion;
* acute coronary syndrome
* congestive heart failure (New York Heart Association (NYHA) classification stage III-IV)
* diabetes mellitus
* chronic kidney disease
* previous PCI in the target vessel
* heavily calcified vessels
* allergy to metformin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-02; Primary Completion 2019-07-31 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Percentage plaque volume change over 24 months | 24 months
  Changes in plaque volume in 24 months

SECONDARY OUTCOMES:
Culprit lesion in-stent restenosis | 24 months
  Neointimal hyperplasia at 24 month follow up
Plaque tissue component percentage change over 24 months | 24 months
  Percentage change in necrotic, fibrotic, lipidic and calcific tissue volume
Correlation of glycemic parameters with plaque characteristics | At index hospitalization and follow up (24 months)
  Correlation of glycemic parameters with plaque characteristics
Plaque volume change in metformin vs non-metformin treated patients over 24 months | 24 months
  Plaque volume change in metformin vs non-metformin treated patients over 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Pauls Stradins Clinical University hospital, Riga, Latvia

IPD SHARING:
Plan to Share IPD: No